CLINICAL TRIAL: NCT05674578
Title: Supporting Black Breast Cancer Survivors: Feasibility Trial of Health Coaching-Based Navigation at the Conclusion of Treatment
Brief Title: Health Coaching-Based Navigation at the Conclusion of Treatment for the Support of Black Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Bridget Oppong, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-21185; NCI-2021-08425 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (patient navigator) (Experimental): Patients are assigned a Black patient navigator for racial concordance and receive coaching from patient navigator over 30 minutes every other week for 3 months and then monthly for 3 months.
  Interventions: Behavioral: Patient Navigation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Patient Navigation — Assigned a patient navigator and receive coaching
  Other Names: Patient Navigator Program
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the feasibility of coaching-based navigation for black breast cancer survivors including recruitment, dropout, and survey completion rates. A coaching-based navigation may perform a needs assessment and coach the participant to access relevant supportive content including physical rehabilitation, emotional and psychosocial support, and nutrition and exercise programming. This trial aims to see whether this navigation program may improve the quality of life of black breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of coaching-based navigation for black breast cancer survivors including recruitment, dropout, and survey completion rates.

SECONDARY OBJECTIVES:

I. To evaluate the preliminary impact of health coaching on completion of scheduled survivorship related referrals and participation in support services.

II. To determine the preliminary impact on quality of life and self-efficacy pre and post coaching.

OUTLINE:

Patients are assigned a Black patient navigator for racial concordance and receive coaching from patient navigator over 30 minutes every other week for 3 months and then monthly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Black women > 18 years of age with stage I-III primary breast cancer who have completed definitive breast cancer treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 6 months
  Will be calculated as the number of new eligible women per month.
Consent rate | Up to 6 months
  Will be calculated as the number of consented women (set to 40 for this study) divided by the total number of women approached.
Dropout rate | Up to 6 months
  Will be calculated as the percentage of women who are enrolled in the study but withdraw before the conclusion of the study.
Patient-Reported Outcomes Measurement Information System score | Up to 6 months
  Differences in scoring at the start of the study period and at the end of the trial will also be summarized by mean, standard deviation, and range.
European Organization for Research and Treatment of Cancer Quality of Life-30 score | Up to 6 months
  Differences in scoring at the start of the study period and at the end of the trial will also be summarized by mean, standard deviation, and range.
Breast Cancer Self Efficacy Scale score | Up to 6 months
  A self reported, unidimensional, 11 item scale designed to show the differences in scoring at the start of the study period and at the end of the trial will also be summarized by mean, standard deviation, and range.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget A Oppong, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT05674578/ICF_000.pdf